CLINICAL TRIAL: NCT00561600
Title: A Randomized, Prospective, Comparative, Multi-Center Clinical Evaluation of the DePuy ASR™-XL Acetabular Cup System vs. the Pinnacle™ Metal- on- Metal Total Hip System Study
Brief Title: Multi-Center Comparative Trial of the ASR™-XL Acetabular Cup System vs. the Pinnacle™ Metal- on- Metal Total Hip System
Acronym: ASR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04062
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-06

CONDITIONS: Non-inflammatory Degenerative Joint Disease
Keywords: Hip arthroplasty; Acetabular cup replacement; Acetabulum arthroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): ASR™-XL Modular Acetabular Cup System stem
  Interventions: Device: ASR™-XL Modular Acetabular Cup System
- B (Active Comparator): Pinnacle™ acetabular shell, with a 28mm or 36mm ULTAMET® metal liner, and a 28mm or 36mm Articul/eze M head.
  Interventions: Device: Pinnacle™ acetabular shell

INTERVENTIONS:
Device: ASR™-XL Modular Acetabular Cup System — The ASR™-XL Modular Acetabular Cup System treatment device is comprised of a metal acetabular cup, a unipolar femoral head and a taper sleeve adapter.
  Other Names: Acetabular cup replacement
  Arms: A
Device: Pinnacle™ acetabular shell — The Pinnacle™ shells are cementless, titanium alloy cups with Porocoat® porous coating and HA DuoFix™ coating. There are various different liners available for use with the Pinnacle™ Acetabular Cup System. For the purpose of this investigation, the CoCrMo ULTAMET® 28mm or 36 mm metal liners will be used.
  Other Names: Acetabular cup replacement
  Arms: B

SUMMARY:
The primary objective of this investigation is to evaluate the clinical and radiographic outcomes of the ASR™-XL Acetabular Cup System compared to the Pinnacle™ Acetabular Cup with a 28mm or 36mm ULTAMET™ metal insert.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to gather sufficient clinical and radiographic data to permit valid scientific comparisons between treatment and control group outcomes. The treatment group/device for this study is the ASR™-XL Acetabular Cup System, and the control group/device is the Pinnacle™ Cup System w/ the 28mm or 36mm ULTAMET™ metal liner. The study objective will be achieved by way of treatment group selection, treatment administration, and management of participating study Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to or capable of providing consent to participate in the clinical investigation.
* Subject is between the ages of 20-75 years, inclusive.
* Subject requires a cementless, primary total hip arthroplasty for non-inflammatory degenerative joint disease (NIDJD).
* Subject has sufficient bone stock for the hip replacement device.
* Subject is a suitable candidate for the devices specified in the clinical investigation plan and is willing to be randomized to either cup system device.

Exclusion Criteria:

* Subject, in the opinion of the Investigator, has an existing condition that would compromise his/her participation and follow-up in this investigation.
* Subject with a known allergy to metal (e.g. jewelry).
* Subject has inflammatory arthritis (e.g. rheumatoid arthritis).
* Subject has active or recent joint sepsis.
* Subject with marked atrophy or deformity in the upper femur.
* Subject with a neuromuscular disease where the loss of musculature would affect functional outcome.
* Subject, in the opinion of the Clinical Investigator, has a history of chronic renal insufficiency (e.g. dialysis).
* Subject is receiving systemic steroid therapy, excluding inhalers or intra-capsular injections, within 3 months prior to surgery.
* Subject with known, active metastatic or neoplastic disease.
* Subject is known to be pregnant, a prisoner, mentally incompetent, and or alcohol or drug abuser.
* Subject is currently involved in any personal injury litigation, medical legal or worker's compensation claims.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Whalen, BS, DC, Study Director — DePuy Orthopaedics
Locations (8):
- United States (8):
  - Desert Orthopaedics, Rancho Mirage, California
  - Resurgens Orthopaedics, Cumming, Georgia
  - Illinois Bone and Joint Institute, Morton Grove, Illinois
  - Spectrum Health Hospital Research, Grand Rapids, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Eastern Oklahoma Orthopedic Center, Tulsa, Oklahoma
  - Orthopaedic Specialists of Austin, Austin, Texas
  - Valley Orthopaedic Associates, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at orthopaedic clinics began Nov 2006 and ended Dec 2009
Groups:
- A ASR™-XL: ASR™-XL Modular Acetabular Cup System stem
- B Pinnacle™: Pinnacle™ acetabular shell, with a 28mm or 36mm ULTAMET® metal liner, and a 28mm or 36mm Articul/eze M head.
Period: Overall Study
Arm/Group | A ASR™-XL | B Pinnacle™
Started | 130 | 135
Completed | 112 | 119
Not Completed | 18 | 16

BASELINE CHARACTERISTICS:
Groups:
- ASR XL: ASR™-XL Acetabular Cup System
- Pinnacle MoM: Pinnacle metal on metal acetabular cup system
- Total: Total of all reporting groups
Arm/Group | ASR XL | Pinnacle MoM | Total
Number analyzed (Participants) | 130 | 135 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.6) | 59.4 (9.4) | 59.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 51 | 111
  Male | 70 | 84 | 154
Region of Enrollment [Number; unit: participants]
  United States | 130 | 135 | 265
BMI [Mean (Standard Deviation); unit: lb/in^2] — Body mass index
  lb/in^2 | 29.7 (7.0) | 30.1 (6.0) | 29.9 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Composite Success Based Upon Harris Hip Score, Radiographic and Survivorship Outcomes
Description: "Composite success: 1) Revision free (life of study) 2) No evidence of radiographic failure (life of study) 3) Harris Hip score => 80 at 24 months"
Time Frame: 24-month interval.
Population: Out of the 265 enrolled subjects, 51 subjects were removed from the analysis for the following reasons: 2 deaths (1 inv, 1 control); 4 protocol violations (0 inv, 4 control); 6 consent withdrawn (2 inv, 4 control); 39 lost to follow-up (17 inv, 22 control).
Measure: Number; unit: participants
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 110 | 104
participants | 82 | 92
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; A non-inferiority test of the proportion successful for each treatment group will be the primary test of efficacy in this investigation. The null hypothesis is Ho: Xc-Xt ≥ 0.08 and the alternative hypothesis is HA:Xc-Xt < 0.08 Sample size of 126 per group was needed assuming 93% success rates, this was increased to 150 per group to account for attrition; Test type: Non-Inferiority or Equivalence — non inferiority of proportion successful with 8% non inferiority margin at 24 months; p = 0.872, Chi-squared; percentage difference = .139, 95% CI 1-sided [upper limit .225] — The upper confidence limit was a priori determined to be a secondary endpoint

2. Secondary Outcome: T-Test of Harris Hip Total Score Means at 24 Months
Description: T-Test of Harris Hip total score means at 24 months
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Units on a scale of 0-100,100 is best.
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 110 | 105
Units on a scale of 0-100,100 is best. | 94.8 (9.4) | 96.4 (6.4)
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; Test type: Superiority or Other; p = 0.167, t-test, 2 sided; Satterthwaite

3. Secondary Outcome: Harris Hip Pain Sub Score at 24 Months
Description: Mean Harris Hip Pain sub score
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on scale of 0-44. 44 is best
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 110 | 106
units on scale of 0-44. 44 is best | 41.5 (6.0) | 42.7 (3.3)

4. Secondary Outcome: Harris Hip Function Score at 24 Months
Description: Mean Harris Hip Function sub score at 24 months
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale 0-47. 47 is best
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 110 | 105
units on a scale 0-47. 47 is best | 31.4 (3.6) | 31.6 (3.7)

5. Secondary Outcome: Analysis of Metal Ion Release - Serum Cobalt
Description: Serum Cobalt
Time Frame: Pre-operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 31 | 32
ug/L | 0.10 [0.07 to 0.18] | 0.10 [0.06 to 0.40]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; Test type: Superiority or Other; p = 0.457, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Analysis of Metal Ion Release - Serum Chromium
Description: Serum Chromium
Time Frame: pre-operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 31 | 32
ug/L | 0.12 [0.07 to 1.30] | 0.12 [0.07 to 2.73]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; Test type: Superiority or Other; p = 0.762, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Cobalt
Description: Erythrocyte cobalt
Time Frame: pre-operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 31 | 32
ug/L | 0.07 [0.05 to 1.26] | 0.08 [0.04 to 0.20]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; Test type: Superiority or Other; p = 0.869, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Chromium
Description: Erythrocyte Chromium
Time Frame: Pre-operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 31 | 32
ug/L | 0.55 [0.20 to 59.45] | 0.62 [0.15 to 2.23]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; Test type: Superiority or Other; p = 0.799, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Analysis of Metal Ion Release - Serum Cobalt
Description: Serum Cobalt
Time Frame: 4 months post-operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 32 | 29
ug/L | 1.39 [0.06 to 10.52] | 0.51 [0.22 to 2.14]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; HO: Pinnacle=ASR-XL. The alternative hypothesis is HA: Pinnacle≠ASR-XL. Serum cobalt ions were expected to be lower in the ASR-XL group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Analysis of Metal Ion Release - Serum Chromium
Description: Serum Chromium
Time Frame: 4 months post operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 32 | 29
ug/L | 1.38 [0.17 to 7.67] | 0.72 [0.25 to 2.48]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; HO: Pinnacle=ASR-XL. The alternative hypothesis is HA: Pinnacle≠ASR-XL. Serum chromium ions were expected to be lower in the ASR-XL group; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Cobalt
Description: Erythrocyte Cobalt
Time Frame: 4 months post-operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 32 | 28
ug/L | 0.85 [0.06 to 8.41] | 0.26 [0.17 to 0.92]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; HO: Pinnacle=ASR-XL. The alternative hypothesis is HA: Pinnacle≠ASR-XL. Erythrocyte cobalt ions were expected to be lower in the ASR-XL group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Chromium
Description: Erythrocyte Chromium
Time Frame: 4 months post-operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 32 | 28
ug/L | 0.45 [0.24 to 11.53] | 0.50 [0.15 to 2.59]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; HO: Pinnacle=ASR-XL. The alternative hypothesis is HA: Pinnacle≠ASR-XL. Erythrocyte chromium ions were expected to be lower in the ASR-XL group; Test type: Superiority or Other; p = 0.882, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Analysis of Metal Ion Release - Serum Cobalt
Description: Serum Cobalt
Time Frame: 12 months post-operative
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL | Pinnacle MoM
Number analyzed (Participants) | 30 | 30
ug/L | 1.55 [0.35 to 25.38] | 0.98 [0.17 to 5.97]
Statistical Analysis 1: Comparison: ASR XL vs Pinnacle MoM; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Analysis of Metal Ion Release - Serum Chromium
Description: Serum Chromium
Time Frame: 12 Months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 30 | 30
ug/L | 1.37 [0.29 to 28.62] | 1.19 [0.39 to 7.19]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.237, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Cobalt
Description: Erythrocyte Cobalt
Time Frame: 12 Months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 30 | 30
ug/L | 0.91 [0.26 to 29.60] | 0.41 [0.14 to 3.56]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Chromium
Description: Erythrocyte Chromium
Time Frame: 12 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 30 | 30
ug/L | 1.12 [0.35 to 22.83] | 0.58 [0.20 to 4.80]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.121, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Analysis of Metal Ion Release - Serum Cobalt
Description: Serum Cobalt
Time Frame: 24 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 25 | 21
ug/L | 3.26 [0.36 to 29.14] | 1.15 [0.22 to 9.39]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Analysis of Metal Ion Release - Serum Chromium
Description: Serum Chromium
Time Frame: 24 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 25 | 21
ug/L | 2.30 [0.32 to 26.67] | 1.48 [0.62 to 7.01]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.103, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Cobalt
Description: Erythrocyte Cobalt
Time Frame: 24 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 25 | 21
ug/L | 1.61 [0.25 to 37.55] | 0.63 [0.20 to 2.70]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Chromium
Description: Erythrocyte Chromium
Time Frame: 24 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 25 | 21
ug/L | 1.29 [0.24 to 7.90] | 1.00 [0.20 to 3.61]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.300, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Analysis of Metal Ion Release - Serum Cobalt
Description: Serum Cobalt
Time Frame: 36 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 30 | 19
ug/L | 3.17 [0.77 to 33.85] | 2.19 [0.36 to 12.63]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.079, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Analysis of Metal Ion Release - Serum Chromium
Description: Serum Chromium
Time Frame: 36 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 30 | 19
ug/L | 1.80 [0.59 to 26.77] | 1.57 [0.27 to 8.73]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.766, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Cobalt
Description: Erythrocyte cobalt
Time Frame: 36 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 30 | 19
ug/L | 2.06 [0.47 to 54.65] | 1.20 [0.26 to 4.74]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.018, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Chromium
Description: Erythrocyte chromium
Time Frame: 36 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 30 | 19
ug/L | 0.76 [0.18 to 7.82] | 0.73 [0.22 to 3.85]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.689, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Analysis of Metal Ion Release - Serum Cobalt
Description: Serum Cobalt
Time Frame: 48 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 15 | 13
ug/L | 3.16 [0.66 to 33.78] | 1.83 [0.46 to 7.37]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.048, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Analysis of Metal Ion Release - Serum Chromium
Description: Serum Chromium
Time Frame: 48 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 15 | 13
ug/L | 2.04 [0.68 to 25.25] | 1.66 [0.36 to 6.04]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.782, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Cobalt
Description: Erythrocyte Cobalt
Time Frame: 48 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 13 | 12
ug/L | 1.90 [0.58 to 40.89] | 1.18 [0.20 to 3.45]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.061, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Analysis of Metal Ion Release - Erythrocyte Chromium
Description: Erythrocyte chromium
Time Frame: 48 months
Population: Metal ion sub-study was limited to two sites. All participants with available data are presented below.
Measure: Median (Full Range); unit: ug/L
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Number analyzed (Participants) | 13 | 12
ug/L | 0.62 [0.21 to 4.21] | 0.62 [0.33 to 1.25]
Statistical Analysis 1: Comparison: ASR XL Acetabular Cup System vs Pinnacle Acetabular Cup System; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.957, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: AE data were collected at 1 month, 4 months, 12 months, 24 months, and annually until study closure. Longest post operative interval with AE data was 60 months.
Arm/Group | ASR XL Acetabular Cup System | Pinnacle Acetabular Cup System
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 72/130 | 59/135
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASR XL Acetabular Cup System (N=130) | Pinnacle Acetabular Cup System (N=135)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Device component issue (General disorders) | 6 (7) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Medical device site reaction (General disorders) | 5 (5) | 1 (1)
Pain (General disorders) | 4 (4) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Infection (Infections and infestations) | 1 (1) | 3 (5)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidacies (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative heterotopic calcification (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 2 (3) | 4 (5)
Blood heavy metal increased (Investigations) | 4 (4) | 0 (0)
Hematocrit decreased (Investigations) | 0 (0) | 1 (1)
White blood cell increased (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (20) | 11 (15)
Arthralgia joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Bone loss (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 12 (19) | 8 (10)
Groin pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (5)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint lock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (11) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotataor cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Piriformis syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Angioplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 5 (6) | 3 (3)
Knee arthroplasty (Surgical and medical procedures) | 2 (3) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Post procedural drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
At study inception, information on whether or not an adverse event was deemed to be serious was not collected. Because of this caveat, the Sponsor has reported all adverse events that occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less